CLINICAL TRIAL: NCT03058796
Title: Contralaterally Controlled FES Plus Video Games for Hand Therapy After Stroke
Brief Title: Contralaterally Controlled Functional Electrical Stimulation Plus Video Games for Hand Therapy After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2249-R; I01RX00249 (Other Grant/Funding Number: Department of Veterans Affairs Rehab. Res. & Dev.)
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Upper Extremity Hemiplegia; Stroke
Keywords: stroke; rehabilitation; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCFES Therapy (Active Comparator): CCFES uses surface electrodes over the paretic finger and thumb extensors to deliver stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove. Thus, volitional opening of the nonparetic hand produces stimulated opening of the paretic hand. CCFES enables stroke survivors to open and close their paretic hand and practice using it in therapy sessions. The treatment regimen includes CCFES-mediated: 1) home-based self-administered hand opening exercises, and 2) lab-based therapist-guided functional task practice.
  Interventions: Device: Contralaterally Controlled Functional Electrical Stimulation (CCFES)
- CCFES Video Game Therapy (Experimental): CCFES Video Game Therapy integrates custom designed hand therapy video games with CCFES which enables participants to use the video game component at home instead of repetitive hand opening exercises.
  Interventions: Device: Contralaterally Controlled Functional Electrical Stimulation (CCFES); Device: Hand Therapy Video Games

INTERVENTIONS:
Device: Contralaterally Controlled Functional Electrical Stimulation (CCFES) — The use of surface electrodes over the paretic finger and thumb extensors to deliver electrical stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove. uses surface electrodes over the paretic finger and thumb extensors to deliver stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove.
  Other Names: CCFES
Device: Hand Therapy Video Games — The use of video games with CCFES to encourage therapeutic hand movement at home
  Other Names: HTVG
  Arms: CCFES Video Game Therapy

SUMMARY:
Determine if adding a video game component to an electrical stimulation therapy improves hand function in stroke patients

DETAILED DESCRIPTION:
A single-blinded randomized controlled trial will be carried out to assess the effects of 12 weeks of Contralaterally Controlled Functional Electrical Stimulation (CCFES) +Hand Therapy Video Games (HTVG) compared to CCFES. Dexterity and activity limitation will be assessed at 0 (baseline), 12 (end of treatment), and 36 (6 months follow-up) wks. The planned treatment dose will be the same for both groups: 10 sessions per week of self-administered treatment at home plus 20 sessions of group-specific occupational therapy in the lab over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

-> 6 months since a first clinical cortical or subcortical, hemorrhagic or nonhemorrhagic stroke

* age 21-80 years old
* unilateral upper limb hemiparesis with finger extensor strength of grade <=4/5 on the Medical Research Council (MRC) scale AND a score of >=1 and <=11/14 on the hand section of the upper extremity Fugl-Meyer Assessment
* adequate active movement of the shoulder and elbow to position the hand in the workspace for table-top task practice (necessary for the lab task practice sessions)
* able to follow 3-stage commands
* able to recall 2 of 3 words after 30 minutes
* surface stimulation of the paretic finger and thumb extensors produces functional hand opening without pain (this will exclude those who have degree of flexor hypertonia that prevents stimulated hand opening)
* Functional passive range of motion (minimal resistance) at elbow, wrist, fingers, and thumb, i.e., there exists enough passive range of motion to reach and acquire table-top objects
* intact vision and hearing
* medically stable
* full voluntary opening/closing of the contralateral (less affected) hand
* demonstrate ability to follow instructions for operating the stimulator or have a caregiver who will assist them

Exclusion Criteria:

* co-existing neurologic diagnosis of peripheral nerve injury, Parkinson's disease, spinal cord injury, traumatic brain injury, or multiple sclerosis
* uncontrolled seizure disorder
* severely impaired cognition and communication
* uncompensated hemineglect
* arm or forearm skin breakdown or edema (to avoid edema-related shunting of current)
* insensate forearm (to avoid risk of electrical burns)
* history of potentially fatal cardiac arrhythmias with hemodynamic instability
* implanted electronic systems (e.g. pacemaker)
* botulinum toxin injections to any upper extremity muscle within 3 months of enrolling
* pregnant women due to unknown risks of surface stimulation during pregnancy
* participating in occupational therapy or other rehabilitation therapies to the upper extremity
* severe shoulder or hand pain

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayme S. Knutson, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knutson JS, Fu MJ, Cunningham DA, Hisel TZ, Friedl AS, Gunzler DD, Plow EB, Busch RM, Pundik S. Contralaterally controlled functional electrical stimulation video game therapy for hand rehabilitation after stroke: a randomized controlled trial. Disabil Rehabil. 2024 Sep;46(19):4466-4475. doi: 10.1080/09638288.2023.2278174. Epub 2023 Nov 14. PMID 37962171

RESULTS

PARTICIPANT FLOW:
Groups:
- CCFES Video Game Therapy: Custom designed hand therapy video games (HTVG) are integrated with CCFES. Surface electrodes over the paretic finger and thumb extensors delivers neuromuscular electrical stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove.
  The therapy regimen includes 12 weeks of CCFES-mediated: 1) home-based self-administered HTVG 10 sessions per week, and 2) lab-based therapist-guided functional task practice 20 sessions over 12 weeks.
- CCFES Therapy: Surface electrodes over the paretic finger and thumb extensors delivers neuromuscular electrical stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove.
  The therapy regimen includes 12 weeks of CCFES-mediated: 1) home-based self-administered hand opening exercises 10 sessions per week, and 2) lab-based therapist-guided functional task practice 20 sessions over 12 weeks.
Period: Overall Study
Arm/Group | CCFES Video Game Therapy | CCFES Therapy
Started | 27 | 25
Completed | 18 | 21
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCFES Video Game Therapy | CCFES Therapy | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 62 (11) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 10 | 22
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Years Since Stroke [Mean (Standard Deviation); unit: years] | 5 (4.5) | 3.9 (3.4) | 4.5 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Box and Block Test Score
Description: The Box and Blocks Test counts how many blocks a patient can pick up, move over a barrier, and release in 60 seconds.
Time Frame: 0 weeks,12 weeks, 36 weeks
Measure: Least Squares Mean (Standard Error); unit: blocks
Arm/Group | CCFES Video Game Therapy | CCFES Therapy
Number analyzed (Participants) | 18 | 21
blocks
  0 weeks | 10.6 (2.6) | 11.0 (2.6)
  12 weeks | 11.2 (2.8) | 12.4 (2.8)
  36 weeks | 11.1 (2.7) | 11.6 (2.6)

2. Secondary Outcome: Action Research Arm Test (ARAT) Score
Description: The ARAT is an activity limitation measure that assesses a subject's ability to handle objects differing in size, weight and shape. Min value = 0 (least functional), Max value = 57 (most functional)
Time Frame: 0 weeks, 12 weeks, 36 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CCFES Video Game Therapy | CCFES Therapy
Number analyzed (Participants) | 18 | 21
units on a scale
  0 weeks | 19.4 (3.6) | 19.0 (2.6)
  12 weeks | 18.6 (3.5) | 21.2 (2.8)
  36 weeks | 18.8 (3.7) | 20.6 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of baseline assessment (0 weeks) until the end of study participation, typically 9 months.
Arm/Group | CCFES Video Game Therapy | CCFES Therapy
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/27 | 2/25
Other Adverse Events (participants affected / at risk) | 8/27 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCFES Video Game Therapy (N=27) | CCFES Therapy (N=25)
Fall leading to hospitalization (Nervous system disorders) | 2 | 1
Car Accident leading to hospitalization (Musculoskeletal and connective tissue disorders) | 1 | 0
Infection leading to hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CCFES Video Game Therapy (N=27) | CCFES Therapy (N=25)
Fall not leading to hospitalization (Nervous system disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT03058796/Prot_SAP_000.pdf